CLINICAL TRIAL: NCT03218371
Title: Scleral Self-indentation During Chandelier-assisted Peripheral Vitrectomy Under Air for Rhegmatogenous Retinal Detachment: A Retrospective Cohort Study.
Brief Title: Scleral Self-indentation Chandelier-assisted Peripheral Vitrectomy Under Air Rhegmatogenous Retinal Detachment.
Status: Completed | Type: Observational
Sponsor: Dar El Oyoun Hospital (Other)
Responsible Party: Principal Investigator, Wael Ahmed Ewais, MD, Lecturer in Department of Ophthalmology, Faculty of Medicine, Cairo University; and consultant vitreoretinal surgeon in Dar El Oyoun Hospital, Dar El Oyoun Hospital
Other Study IDs: DEO00001258
Record Dates: First submitted 2017-07-07; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Retinal Detachment
Keywords: scleral indentation; chandelier light; air vitrectomy; rhegmatogenous retinal detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group (Indentation): Eyes (participants) for whom chandelier-assisted peripheral vitrectomy under air had been performed with scleral indentation. (Exposure)
  Interventions: Procedure: chandelier-assisted peripheral vitrectomy under air
- control group (Non-indentation): eyes (participants) for whom chandelier-assisted peripheral vitrectomy under air had been performed without scleral indentation.
  Interventions: Procedure: chandelier-assisted peripheral vitrectomy under air

INTERVENTIONS:
Procedure: chandelier-assisted peripheral vitrectomy under air — chandelier-assisted peripheral vitrectomy under air for management of peripheral vitreous during RD vitrectomy; whether using indentation or non-indentation

SUMMARY:
The investigators compared the incidence of trimming-induced retinal breaks, retinal redetachment rate, and final LogMAR BCVA; between scleral self-indentation and non-indentation during chandelier-assisted peripheral vitrectomy under air for eyes with primary retinal detachment. Self-indentation enables complete trimming of the vitreous base without causing iatrogenic retinal breaks, with a higher retinal reattachment rate, and with less need for chandelier shift than with non-indentation approach.

DETAILED DESCRIPTION:
Retrospective cohort study. One hundred and thirty eyes of 130 participants with primary rhegmatogenous retinal detachment were identified. All the participants had undergone a chandelier-assisted peripheral vitrectomy under air. Scleral self-indentation had been used in 68 eyes (study group) (Indentation group), while non-indentation had been used in 62 eyes (comparison group) (Non-indentation group). Outcome variables included: Trimming-induced retinal breaks (TIRB), retinal redetachment rate, final LogMAR BCVA, and intraoperative complications.

ELIGIBILITY:
Inclusion Criteria:

- RRD with postoperative follow up > 3 months, without PVR, or with PVR A-B

Exclusion Criteria:

* RRD with less than 3 months of postoperative follow-up,
* RRD with proliferative vitreoretinopathy grade C (PVR C),
* RRD with uveitis,
* RRD with choroidal detachment,
* Giant retinal tears,
* Retinal dialysis,
* Myopic macular hole RRD,
* Traumatic RD,
* Children < 16 years old,
* The later vitrectomy (if vitrectomy had been performed for RRD in both eyes)

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a retrospective cohort study that was done on eyes (participants) with rhegmatogenous retinal detachment (RRD) for whom chandelier-assisted peripheral vitrectomy under air (CPVA) had been performed; whether using scleral self-indentation (Exposure), or without scleral self-indentation (control)
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Trimming-induced retinal breaks (TIRB) (yes/ No) | intraoperative
  number of eyes with iatrogenic retinal breaks along vitreous base during vitreous base trimming

SECONDARY OUTCOMES:
number of Trimming-induced retinal breaks (TIRB) | intraoperative
  number of iatrogenic retinal breaks along vitreous base during vitreous base trimming
retinal redetachment rate (yes/no) | within 3 months
  number of eyes in which recurrent retinal detachment occurred
final LogMAR BCVA | final follow-up visit ( at least 3 months)
  best spectacle corrected visual acuity measured by decimal charts then converted to LogMAR
snellen BCVA > 20/100 (yes/ no) | 3 months
  number of eyes with best corrected visual acuity better than snellen's 20/100 measured by snellen's chart
Chandelier shift (yes/no) | intraoperative
  the need to shift position of chandelier light
Local anaesthesia augmentation (yes/no) | intraoperative
  the need for augmenting local anesthesia for the participant to tolerate indentation

CONTACTS AND LOCATIONS:
Overall Officials: Wael A Ewais, MD, Principal Investigator — consultant vitreoretinal surgeon
Locations (1):
- Dareloyoun hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No